CLINICAL TRIAL: NCT05630963
Title: Beyond Monoamines: The Role of the Nociceptin/Orphanin FQ Receptor in Major Depression
Status: Recruiting | Type: Observational
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Diego Pizzagalli, Director, Center for Depression, Anxiety and Stress Research, Mclean Hospital
Other Study IDs: 2018P000318; 4R37MH068376-17 (NIH)
Record Dates: First submitted 2022-11-16; First posted 2022-11-30 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples are collected seven times over the course of the MRI visit to be assayed for salivary cortisol
  Blood samples are collected during the MRI visit-once before the scan and once after the scan-to processed for RNA, DNA, and serum. Processed samples will be analyzed for proinflammatory cytokines and transcription control levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- MDD subjects: Subjects diagnosed with Major Depression Disorder
  Interventions: Device: Aversive stimuli; Drug: PET radiotracer
- Remitted MDD subjects: Subjects with a history of major depressive disorder episode in the past
  Interventions: Device: Aversive stimuli; Drug: PET radiotracer
- Control subjects: Subjects with no history of known neurological and psychiatric illness.
  Interventions: Device: Aversive stimuli; Drug: PET radiotracer

INTERVENTIONS:
Device: Aversive stimuli — Electrotactile stimulation will be used as the aversive stimulus. The aversive stimulus is delivered in the form of a mild half-second stimulation to the ankle, calibrated to a subjective threshold that is uncomfortable but not painful. This stimulation is delivered by Digitimer DS8R Constant Current Stimulator (Digitimer North America, LLC. Ft. Lauderdale, FL). Its previous model DS71 has been safely implemented in studies with previously MGH-approved IRB's (Milad et al., 2013).
Drug: PET radiotracer — A Nociceptin/Orphanin FQ ("N/OFQ") peptide tracer ([11C] NOP-1A) will be used as the PET radiotracer. Approximately 10 mCi of this tracer will be delivered intravenously as a slow bolus over 60 seconds with beginning of the PET imaging acquisition. Approximately 60 ml of blood will be drawn from an artery throughout the dynamic PET acquisition in order to measure the blood N/OFQ levels.

SUMMARY:
This study looks at the role of the Nociceptin/Orphanin FQ receptor system in the brain of individuals with current or past major depressive disorder (MDD). It also examines how individuals with a history of depression make certain decisions and which brain regions are involved in such decisions. Information collected through MRI, PET, biospecimens (i.e., blood, saliva) and behavioral tasks will be used to predict depressive symptoms in the future.

DETAILED DESCRIPTION:
The overarching goals of this research are to investigate: (1) the activity of the Nociceptin/Orphanin FQ receptor system among individuals with current or remitted MDD; (2) neural foundations of approach/avoidance behaviors in current or remitted MDDs; (3) stress-induced inflammation in individuals with remitted MDD; (4) neural markers that predict future disease course.

This will be achieved through an innovative method of using functional magnetic resonance imaging (fMRI) during an approach/avoidance decision-making task, in addition to a resting positron emission tomography (PET) scan.

ELIGIBILITY:
Inclusion Criteria for all participants:

* All genders, races, and ethnic origins, aged between 18 and 45
* Capable of providing written informed consent, and fluent in English
* Right-handed
* Absence of any psychotropic medications for at least 2 weeks
* Has a smartphone (iPhone or Android) (needed for Ecological Momentary Assessment)

Inclusion Criteria for "Remitted MDD" group:

* Meets inclusion criteria for all subjects, plus:
* History of MDD as defined by DSM-5
* Absence of anxiety disorder for the past two months

Inclusion Criteria for "Current MDD" group:

* Meets inclusion criteria for all subjects, plus:
* Presence of MDD as defined by DSM-5
* Absence of anxiety disorder for the past two months

Exclusion Criteria for all participants:

* Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician. These patients will be immediately referred to appropriate clinical treatment
* Pregnant women or women of childbearing potential who are not using a medically accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, spermicide, IUD, s/p tubal ligation, or partner with vasectomy)
* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* History of seizure disorder
* History of psychiatric illnesses, other than depression or anxiety disorders among the Current MDD and Remitted MDD groups
* History of substance use disorder or alcohol use disorder (as these terms are defined by DSM-5); except depressed subjects may have a history of 'Mild' substance/alcohol use disorder only if it ended as least 12 months ago
* History of cocaine or stimulant use or dopaminergic drugs
* History or current diagnosis of dementia, or a score of < 26 on the Mini Mental State Examination at the screening visit;
* Patients with mood congruent or mood incongruent psychotic features
* Current use of other psychotropic drugs
* Clinical or laboratory evidence of hypothyroidism
* Patients with a lifetime history of electroconvulsive therapy (ECT)
* Failure to meet standard MRI safety requirements
* Abnormal ECG and lab results
* History of seizure disorder
* Contraindications for arterial line (e.g., abnormal result on Allen test, Raynaud's syndrome, history of anemia or bleeding disorder, history of fainting from blood draws).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subjects for this research will be 228 participants recruited from the community by the Center for Depression, Anxiety and Stress Research (Director: Dr. Diego Pizzagalli, Ph.D.). Demographically-matched participants will include: (1) 38 participants with current MDD; (2) 38 participants with past MDD; and (3) 38 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical Interview | Baseline
  For assessing psychological state
Behavioral Performance on the Probabilistic Reward Task (PRT) | Baseline
  the PRT assesses individuals' ability to learn from rewards
MRI Data | within 30 days of Screening Visit
  For testing the neural correlates of approach-avoidance decision making behaviors
Salivary Cortisol | Baseline
  For assessing stress level
PET Data | within 30 days of Screening Visit
  For assessing the Nociceptin/Oprhanin FQ receptor system activity
Arterial blood data | Baseline
  for PET modeling and assessing Nociceptin/Orphanin FQ levels in bloodstream
Follow-up Clinical Interviews | Change from Baseline at 6 months and 12 months after the PET visit
  To assess psychological state changes

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI) | Change from Baseline at 6 months and 12 months after the PET visit
  self-report measure of depressive symptoms
Childhood Trauma Questionnaire (CTQ) | Baseline
  self-report measure of childhood trauma
Medical Outcome Survey-Short form (SF-36) | Change from Baseline at 6 months and 12 months after the PET visit
  self-report with subscales measuring physical functioning, physical role functioning, social functioning, etc.
Perceived Stress Scale (PSS) | Change from Baseline at 6 months and 12 months after the PET visit
  self-report measure of stress levels
Positive and Negative Affect Schedule (PANAS) | Baseline
  self-report measure of positive and negative affect
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | Change from Baseline at 6 months and 12 months after the PET visit
  self-report measure of satisfaction and enjoyment across domains (e.g., work, leisure, social relations)
Snaith Hamilton Pleasure Scale (SHAPS) | Change from Baseline at 6 months and 12 months after the PET visit
  self-report measure of pleasure
Thought and Feeling Questionnaire (TFQ) | Baseline
  self-report measure of perception of being stuck in difficult situations
Defeat Scale (DS) | Baseline
  self-report measure of perception of defeat
Questionnaire of Unpredictability in Childhood (QUIC) | Change from Baseline at 6 months and 12 months after the PET visit
  self-report measure of unpredictability of parental environment growing up
Mood and Anxiety Symptom Questionnaire (MASQ) | Baseline
  self-report measure of mood symptom severity including 4 subscales related to depression and anxiety
State-Trait Anxiety Inventory (STAI) | Baseline
  Measures and differentiates between anxiety
PRT Post-task Questionnaire | Baseline
  self-report measure of participants' thoughts regarding the PRT task stimuli
Temporal Experience of Pleasure Scale (TEPS) | Change from Baseline at 6 months and 12 months after the PET visit
  self-report measure of ability to want and enjoy rewards
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline
  clinical measure of suicidality
Hamilton-Depression Rating Scale (HAMD-17) | Change from Baseline at 6 months and 12 months after the PET visit
  clinical measure of depression severity
Quick Inventory of Depressive Symptomatology (QIDS) | Change from Baseline at 6 months and 12 months after the PET visit
  clinical measure of depression severity
Cognitive-Behavioral Avoidance Scale (CBAS) | Baseline
  self-report measure of trait avoidance
Stress and Adversity Inventory (STRAIN) | Change from Baseline at 12 months after the PET visit
  self-report measure of lifetime exposure to acute and chronic stress that may affect mental and physical health

CONTACTS AND LOCATIONS:
Overall Officials: Diego Pizzagalli, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided